CLINICAL TRIAL: NCT00413933
Title: Comprehensive Intervention for Falls Prevention in the Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of funding
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Yan Press, head of Unit for Community Geriatrics, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sor444506ctil
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2006-12

CONDITIONS: Accidental Falls
Keywords: falls; prevention; elderly; multidisciplinary intervention; health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

ARMS (2):
- Intrevention group (Experimental): each subject in intervention group will get 15 weekly sessions (each session - 45 minutes) of specified exercise from a physical therapist that specializes in fall prevention and walking device recommendations. All subjects will get brochure for home exercise. It will be expected for intervention group to exercise twice daily, each time for 20 minutes in addition to the PT sessions
  Interventions: Procedure: Comprehensive Multidisciplinary Intervention
- Control group (No Intervention): Those who agree to participate in the study will fill in questionnaire about falls (causes, circumstance, results). All will pass through: cognitive assessment by the Mini-Mental State Examination (MMSE), affective assessment by the 15-item Geriatric Depression Scale (GDS), functional assessment by Barthel Index (BI), visual assessment by Snellen charts and basic gait assessment by a "Timed get Up and Go" test (TU&G).
  Participants that fulfill inclusion criteria will be randomly assigned to the intervention group or the control group

INTERVENTIONS:
Procedure: Comprehensive Multidisciplinary Intervention — Comprehensive Multidisciplinary Intervention
  Arms: Intrevention group

SUMMARY:
The purpose of this study is to determine whether the comprehensive multidisciplinary intervention (geriatrician, physical therapist and occupational therapist falls risk assessment and intervention)is effective in the falls prevention in the community dwelling elderly.

DETAILED DESCRIPTION:
Falls and related injuries among elderly people are a major public health problem worldwide.All older people with recurrent falls or assessed as being at increased risk of falling should be considered for an individualized multifactorial intervention.

In successful multifactorial intervention programmes the following specific components are common - against a background of the general diagnosis and management of causes and recognized risk factors:

* exercise
* home hazard assessment and intervention
* vision assessment and referral
* medications list review with modification/withdrawal We will address to 4000 randomly chosen patients from study population (elderly (65+) men and women, living in Beer-Sheva and Ofakim , Israel and belonging to Clalit HMO). This telephone interview will be conducted to reveal falls in last 12 months. The people who do fall (1 + falls) will be invited to research assistant.

In that meeting the research assistant will explain about the study aims and ask them to sign informed consent. Those who do not agree to participate - will be referred to their family doctor for further assessment.

Those who agree to participate in the study will fill in questionnaire about falls (causes, circumstance, results). All will pass through: cognitive assessment by the Mini-Mental State Examination (MMSE), affective assessment by the 15-item Geriatric Depression Scale (GDS), functional assessment by Barthel Index (BI), visual assessment by Snellen charts and basic gait assessment by a "Timed get Up and Go" test (TU&G).

Participants that fulfill inclusion criteria will be randomly assigned to the intervention group or the control group. All participants will be instructed to call to the research assistant closely to each fall.

All information about assessment of patients in both groups will be transferred to the family physician. Their family physician according to his opinion will treat patients from usual care group.

A geriatrician, physiotherapist and occupational therapist will observe patients in the intervention group. OT will conduct a home visit to assess hazard and level of risk factor for falling. Results of assessment will be discussed on multi- disciplinary team meeting.

According to this plan each patient in this group will receive one or more following interventions:

1. Written recommendation to the family physician for medication adjustment. As well, the geriatrician will discuss with family physician these recommendations.
2. Recommendation to the family physician to refer the patient to optometrist/ ophthalmologist.
3. Physical therapy: each subject in intervention group will get 15 weekly sessions (each session - 45 minutes) of specified exercise from a physical therapist that specializes in fall prevention and walking device recommendations. All subjects will get brochure for home exercise. It will be expected for intervention group to exercise twice daily, each time for 20 minutes in addition to the PT sessions.
4. Occupational therapy: OT will make recommendation for changing any unsafe environments in the home.

First follow-up (four months after baseline assessment):

1. OT will make a second home visit to each subject of the intervention group to check recommendation fulfillment.
2. Study assistant will repeat baseline assessment (MMSE, GDS, BI, TU&G and visual assessment by Snellen chart).
3. Information about falls and injuries as well as health care utilization will be collected from Clalit computerized system and Soroka Medical Center data base.
4. Information about medication adjustment and changes will be collected from Clalit computerized system.

Second follow-up (12 months after baseline assessment ) :

1. Study assistant will repeat baseline assessment (MMSE, GDS, BI, TUG test and visual assessment by Snellen chart).
2. Information about falls and injuries as well as health care utilization will be collected from Clalit computerized system and Soroka Medical Center data base.
3. Information about medication adjustment and changes will be collected from Clalit computerized system.

ELIGIBILITY:
Inclusion Criteria:

* Living in Beer Sheva or Ofakim , Israel
* Members of Clalit HMO
* 1 or more falls in past 12 month (self-reported)
* Age 65 or more
* Mobile outdoors without wheelchair

Exclusion Criteria:

* Seriously ill patients - as dyspnea with light exercise, unstable heart disease
* MMSE less than 18

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
number of falls | 4 and 12 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Yan Press, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Department of Family Medicine, Faculty of Health Sciences, Ben Gurion University of the Negev, Beersheba, Israel